CLINICAL TRIAL: NCT05652647
Title: A PHASE 1, OPEN-LABEL, 2-PERIOD, FIXED SEQUENCE STUDY TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM AND EXCRETION OF [14C]PF-07081532 AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-07081532 IN HEALTHY MALE PARTICIPANTS USING A [14C]-MICROTRACER APPROACH
Brief Title: A Study to Understand How the Study Medicine (PF-07081532) is Processed and Eliminated in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3991006
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy Participants
Keywords: Absorption; Distribution; Metabolism; Elimination; Bioavailability; Fraction absorbed; Mass balance; Healthy Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- One group of healthy adult male participants (Experimental)
  Interventions: Drug: Oral [14C]PF-07081532; Drug: Oral PF-07081532 and IV [14C]PF-07081532

INTERVENTIONS:
Drug: Oral [14C]PF-07081532 — A single oral dose of [14C]PF-07081532, will be administered as a liquid formulation in study period 1.
Drug: Oral PF-07081532 and IV [14C]PF-07081532 — In study period 2: a single, oral, unlabeled dose of PF-07081532 will be administered as a liquid formulation. Approximately 1 hours after the administration of the unlabeled oral dose, a single dose of [14C]PF-07081532 will be administered via intravenous infusion.

SUMMARY:
The purpose of this clinical trial is to learn about how much PF-07081532 will be taken up and processed by healthy male participants. The study consists of two parts, called study periods. In Period 1, participants will take one dose of PF-07081532 by mouth. In Period 2, participants will take one dose by mouth and one dose as an injection through a vein at the study clinic.

In Period 1, participants will stay at the clinic site for up to 21 days. In Period 2, they will stay at the clinic site for 7 days. During their stays, participants will have their blood, urine, and feces collected by the study doctors several times. We will measure the level of PF-07081532 in participants' blood, urine, and feces samples. This will help us know how much the study medicine is getting taken in by the body. At the end of the study, participants will be contacted by phone to check in. Participants will be involved in this study for about 12 weeks.

ELIGIBILITY:
Key Eligibility criteria for this study include, but are not limited to the following:

Inclusion criteria:

Healthy Male participants must be 18 to 60 years of age, inclusive.

Overtly healthy as determined by medical evaluation including medical history, physical examination, blood pressure and pulse rate measurement, standard 12-lead ECG, and laboratory tests.

BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion criteria:

History of irregular bowel movements (eg, irritable bowel syndrome, frequent episodes of diarrhea, or constipation defined by less than 1 bowel movement on average per 2 days) or lactose intolerance

Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).

Previous administration with an investigational product (drug or vaccine) within 90 days (or as determined by the local requirement) preceding the first dose of study intervention used in this study.

Total 14C radioactivity measured in plasma exceeding 11 mBq/mL.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 6 participants were enrolled and treated in both Period 1 and Period 2 of the study.
Groups:
- Period 1: [14C]PF-07081532 30 mg Oral; Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV: In Period 1, participants received a single oral dose of [14C]PF-07081532 30 mg; in Period 2, participants received an oral dose of unlabeled PF-07081532 30 mg, followed by intravenous (IV) infusion of [14C]PF-07081532 100 µg.
Period: Overall Study
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral; Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled and treated.
Groups:
- Period 1: [14C]PF-07081532 30 mg Oral; Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV: In Period 1, participants received a single oral dose of [14C]PF-07081532 30 mg; in Period 2, participants received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg.
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral; Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-25 years | 0
  26-35 years | 5
  36-45 years | 0
  >45 years | 1
Age, Customized [Median (Full Range); unit: Years] | 32 [29 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Recovery of Radioactivity in Urine, Feces and Both Routes Combined, as Percentage of Orally Administered Radioactive Dose of [14C]PF-07081532
Description: Urine and feces samples collected after a single oral dose of [14C]PF-07081532 30 mg (~250 nCi) in Period 1 were analyzed using Accelerator Mass Spectrometry (AMS). "Blank" pre-dose urine samples were collected within the 24 hours prior to dosing, "blank" fecal samples were collected from at least 1 bowel movement within the 48 hours prior to dosing. Following oral dosing, each urine void was collected across intervals of 0-12 hours, 12-24 hours, and each subsequent 24 hour interval up to 360 hours post dose, and all feces excreted were collected across each 24 hour interval up to 360 hours post dose. Recovery of radioactivity in urine, feces, and both routes combined, determined as percentage of the orally administered radioactive dose, are reported.
Time Frame: 360 hours
Population: The analysis population included all evaluable participants who had received 1 dose of [14C]PF-07081532 in Period 1 with complete total radioactivity concentration (urinary and fecal) data and who had no protocol deviations that might have affected the extent of excretion analysis.
Measure: Mean (Standard Deviation); unit: Percentage of radioactive dose
Groups:
- Period 1: [14C]PF-07081532 30 mg Oral: In Period 1, participants received a single oral dose of [14C]PF-07081532 30 mg.
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
Percentage of radioactive dose
  Urine | 4.7 (0.6)
  Feces | 78.6 (6.7)
  Urine + Feces | 83.4 (6.9)

2. Primary Outcome: Relative Abundance of [14C]PF-07081532 and Its Metabolites in Plasma After A Single Oral Dose of [14]PF-07081532 in Period 1
Description: Plasma samples collected after a single oral dose of [14C]PF-07081532 30 mg (~250 nCi) were analyzed using Ultra Performance Liquid Chromatography coupled to High Resolution Mass Spectrometry (UPLC-HRMS). Relative abundance = (sum of radioactive content of fractions contributing to a particular peak/total circulating drug-related material [total [14C] radioactivity in plasma]) x 100%. Metabolites that were detected and identifiable (including coeluting metabolites reported together) are reported in this outcome measure (OM).
Time Frame: Pre-dose (0 hours [hrs]) and 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 6 hrs, 8 hrs, 10 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs, and 72 hrs post Period 1 Day 1 dosing
Population: The analysis population included all participants who received study intervention of [14C]PF-07081532 in Period 1.
Measure: Number; unit: Percentage of circulating radioactivity
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
Percentage of circulating radioactivity
  767a (hydroxy glucuronide) | 1.2
  PF-07943285 (hydroxy glucuronide) | 8.8
  767c (hydroxy glucuronide) | 0.4
  671 (hydroxy sulfate) | 0.6
  Coeluting components: PF-07214855, PF-07260051, PF-07943284 | 9.1
  PF-07081532 | 79.3
  Unassigned [14C] | 0.6

3. Primary Outcome: Relative Abundance of [14C]PF-07081532 and Its Metabolites in Urine and Feces After A Single Oral Dose of [14]PF-07081532 in Period 1
Description: Urine and feces samples collected after a single oral dose of [14C]PF-07081532 30 mg (~250 nCi) were analyzed using UPLC-HRMS. "Blank" pre-dose urine samples were collected within the 24 hours prior to dosing, "blank" fecal samples were collected from at least 1 bowel movement within the 48 hours prior to dosing. To obtain samples for evaluation of relative abundance in urine and feces, following oral dosing, each urine void was collected across intervals of 0-12 hours, 12-24 hours, and each subsequent 24 hour interval up to 96 hours post dose, and all feces excreted were collected across each 24 hour interval up to 144 hours post dose. Relative abundance was determined as sum of radioactive content of fractions contributing to a particular peak divided by total radioactive dose excreted in urine/feces respectively. Metabolites that were detected and identifiable (including coeluting metabolites reported together) are reported in this OM.
Time Frame: 96 hours for urine samples and 144 hours for feces samples
Population: The analysis population included all participants who received study intervention of [14C]PF-07081532 in Period 1.
Measure: Number; unit: Percentage of radioactive dose
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
Percentage of radioactive dose
  Urine: PF-07943285 (hydroxy glucuronide) | 0.1
  Urine: 767c (hydroxy glucuronide) | 0.03
  Urine: coeluting components PF-07214855 , PF-07260051 and PF-07943284 | 0.2
  Urine: PF-07081532 | 0.04
  Urine: Unassigned [14C] | 4.33
  Feces: PF-07240437 (catechol) | 3.89
  Feces: PF-07943283 (hydroxy) | 13.6
  Feces: coeluting components PF-07260051 and PF-07943284 | 24.7
  Feces: PF-07081532 | 13.2
  Feces: Unassigned [14C] | 23.2

4. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Total [14C] After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration of total [14C] after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1. AUC for total [14C] is presented as nanogram equivalent * hour/milliliter (ngEq*hr/mL).
Time Frame: Pre-dose (0 hrs) and 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 6 hrs, 8 hrs, 10 hrs, 12 hrs, 15 hrs, 24 hrs, 36 hrs, 48 hrs, 72 hrs, 96 hrs, 120 hrs and 144 hrs post Period 1 Day 1 dosing
Population: The analysis population included all participants dosed with [14C]PF-07081532 in Period 1 who had at least one of the PF-07081532 or total [14C] PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
ngEq*hr/mL | 74360 (17)

5. Secondary Outcome: AUClast of PF-07081532 After A Single Oral Dose of [14]PF-07081532 in Period 1
Description: Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration of PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hr/milliliter (ng*hr/mL)
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
nanogram*hr/milliliter (ng*hr/mL) | 49380 (21)

6. Secondary Outcome: Plasma Maximum Observed Concentration (Cmax) of Total [14C] After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Maximum plasma concentration of total [14C] after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent/milliliter (ngEq/mL)
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
nanogram equivalent/milliliter (ngEq/mL) | 2934 (10)

7. Secondary Outcome: Plasma Cmax of PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Maximum plasma concentration of PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
nanogram/milliliter (ng/mL) | 2874 (10)

8. Secondary Outcome: Plasma Time to Reach Cmax (Tmax) of Total [14C] and PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Time to reach maximum plasma concentration of total [14C] and PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
hour
  Total [14C] | 4.93 [2.00 to 6.00]
  PF-07081532 | 3.93 [2.00 to 6.00]

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve to Infinity (AUCinf) of Total [14C] After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Area under the plasma concentration versus time curve from time zero to infinity of total [14C] after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
ngEq*hr/mL | 76050 (17)

10. Secondary Outcome: AUCinf of PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Area under the plasma concentration versus time curve from time zero to infinity of PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
ng*hr/mL | 51370 (21)

11. Secondary Outcome: Plasma Elimination Half Life (t1/2) of Total [14C] and PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Plasma elimination half-life of total [14C] and PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
hour
  Total [14C] | 65.20 (6.7308)
  PF-07081532 | 19.42 (3.5583)

12. Secondary Outcome: Apparent Clearance of Drug From Plasma (CL/F) of PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Apparent clearance of PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F was calculated as dose/AUCinf, where AUCinf was area under the plasma concentration versus time curve from time zero to infinity.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
Liter/hour (L/hr) | 0.5851 (22)

13. Secondary Outcome: Plasma Apparent Volume of Distribution (Vz/F) of PF-07081532 After A Single Oral Dose of [14C]PF-07081532 in Period 1
Description: Apparent volume of distribution of PF-07081532 after the participant received a single oral dose of [14C]PF-07081532 30 mg (approximately 250 nCi [14C]) in Period 1. Vz/F is calculated as Dose/(AUCinf * kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve, AUCinf is area under the plasma concentration versus time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral
Number analyzed (Participants) | 6
L | 16.13 (21)

14. Secondary Outcome: Plasma AUClast of [14C]PF-07081532 Following Intravenous (IV) Administration of [14C]PF-07081532 in Period 2
Description: Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration of [14C]PF-07081532 after the participant received an oral (PO) dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose).
Time Frame: Pre-dose (0 hrs) and 0.17 hrs, 0.25 hrs, 0.33 hrs, 0.5 hrs, 1 hr, 3 hrs, 5 hrs, 7 hrs, 9 hrs, 11 hrs, 14 hrs, 23 hrs, 35 hrs, 47 hrs, 71 hrs, 95 hrs, 119 hrs and 143 hrs post IV dosing of [14C]PF-07081532 on Period 2 Day 1
Population: The analysis population included all participants dosed with [14C]PF-07081532 in Period 2 who had at least one of the [14C]PF-07081532 PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV: In Period 2, participants received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg.
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng*hr/mL | 185.9 (32)

15. Secondary Outcome: Dose-Normalized Plasma AUClast (AUClast(dn) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Dose-normalized plasma AUClast of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (equivalent to 0.1 mg; approximately 1 hour after the oral dose). AUClast(dn) = AUClast/Dose, where AUClast = area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration, dose = IV dose of [14C]PF-07081532 (expressed in mg).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng*hr/mL/mg | 1831 (28)

16. Secondary Outcome: Plasma Cmax of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Maximum plasma concentration of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng/mL | 23.20 (16)

17. Secondary Outcome: Dose-Normalized Plasma Cmax (Cmax (dn)) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Dose-normalized plasma Cmax of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (equivalent to 0.1 mg; approximately 1 hour after the oral dose). Cmax(dn) = Cmax/Dose, where Cmax = maximum concentration, dose = IV dose of [14C]PF-07081532 (expressed in mg).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng/mL/mg | 228.5 (13)

18. Secondary Outcome: Plasma Tmax of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Time to reach maximum plasma concentration of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
hour | 0.250 [0.250 to 0.267]

19. Secondary Outcome: Plasma AUCinf of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Area under the plasma concentration versus time curve from time zero to infinity of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng*hr/mL | 186.9 (32)

20. Secondary Outcome: Dose-Normalized Plasma AUCinf (AUCinf(dn)) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Dose-normalized plasma AUCinf of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (equivalent to 0.1 mg; approximately 1 hour after the oral dose). AUCinf(dn) = AUCinf/Dose, where AUCinf = area under the plasma concentration versus time curve from time zero to infinity, dose = IV dose of [14C]PF-07081532 (expressed in mg).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
ng*hr/mL/mg | 1844 (29)

21. Secondary Outcome: Plasma t1/2 of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Plasma terminal half life of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
hour | 21.02 (2.9027)

22. Secondary Outcome: Plasma Clearance (CL) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Plasma clearance of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose). Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL was calculated as (IV dose of [14C]PF-07081532) divided by (AUCinf of [14C]PF-07081532), where AUCinf = Area under the plasma concentration versus time curve from time zero to infinity.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
L/hr | 0.5420 (29)

23. Secondary Outcome: Plasma Steady-State Volume of Distribution (Vss) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Plasma steady-state volume of distribution of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose). Vss was calculated as CL * MRT, where CL was the plasma clearance of [14C]PF-07081532, and MRT was the Mean Residence Time of [14C]PF-07081532. MRT = AUMCinf/AUCinf - (Infusion time/2), where AUMCinf was the area under the first moment curve from time zero to infinity, AUCinf = area under the plasma concentration versus time curve from time zero to infinity.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
L | 10.70 (15)

24. Secondary Outcome: Plasma Mean Residence Time (MRT) of [14C]PF-07081532 Following IV Administration of [14C]PF-07081532 in Period 2
Description: Plasma mean residence time of [14C]PF-07081532 after the participant received an oral dose of unlabeled PF-07081532 30 mg, followed by IV infusion of [14C]PF-07081532 100 µg (approximately 1 hour after the oral dose). MRT = AUMCinf/AUCinf - (Infusion time/2), where AUMCinf was the area under the first moment curve from time zero to infinity, AUCinf = area under the plasma concentration versus time curve from time zero to infinity.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
hour | 19.77 (21)

25. Secondary Outcome: Absolute Oral Bioavailability (F) of PF-07081532 in Period 2
Description: F is a measure of the rate and extent of a drug reaching the systemic circulation in its unchanged form. F was estimated as the ratio of adjusted geometric means of dose-normalized plasma AUCinf following oral unlabeled PF-07081532 and IV [14C]PF-07081532 in Period 2, which is equivalent to the following equation: F = (AUCpo/[14C]_AUCiv)*([14C]_Doseiv/Dosepo). AUCpo and [14C]_AUCiv were the AUCinf values of unlabeled PF-07081532 and [14C]PF-07081532, respectively in Period 2; Dosepo and [14C]_Doseiv were the 30 mg oral dose of unlabeled PF-07081532 and each participant's individual IV dose of [14C]PF-07081532, respectively.
Time Frame: Pre-dose (0 hrs) and 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 6 hrs, 8 hrs, 10 hrs, 12 hrs, 15 hrs, 24 hrs, 36 hrs, 48 hrs, 72hrs, 96 hrs, 120 hrs and 144 hrs post oral dosing of unlabeled PF-07081532 on Period 2 Day 1
Population: The analysis population included all participants dosed with PF-07081532 and [14C]PF-07081532 in Period 2 who had at least one of the PK parameters of interest.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent
Arm/Group | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
Percent | 90.79 [84.62 to 97.41]

26. Secondary Outcome: Fraction Absorbed (Fa) of PF-07081532
Description: Fa was estimated as the ratio of adjusted geometric means of the % of administered radioactive dose excreted into urine following oral (Period 1) and IV (Period 2) dosing of [14C]PF-07081532. Urine radioactivity up to Day 7 in Period 1 was used to match the duration of Period 2 urine collection. Fa = (Total [14C]_Urine_PO_Trunc/Total [14C]_Urine_IV) × ([14C] Doseiv/[14C] Dosepo). Total [14C]_Urine_PO_Trunc = Total cumulative radioactivity excreted into urine from time zero up to Day 7 following Period 1 oral dosing, calculated as sum of ([14C] urine concentration × sample volume) for each collection interval. Total [14C]_Urine_IV = Total cumulative radioactivity excreted into urine from time zero to the time of last measurable concentration following Period 2 IV dosing, calculated as sum of ([14C] concentration × urine collection volume) for each collection interval (= sum of collection intervals). [14C] Dose = radioactivity dose (PO in Period 1, IV in Period 2) for each participant.
Time Frame: Day 1 to Day 7 for both Period 1 and Period 2
Population: The analysis population included all participants who received at least 1 dose of study intervention and had at least 1 of the PF-07081532 or [14C]PF-07081532 parameters of interest.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral; Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6
Percent | 79.91 [73.53 to 86.85]

27. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. TEAEs were AEs that occurred after initiation of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect.
Time Frame: Maximum of 11 weeks
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6 | 6
Participants
  All-causality TEAE | 4 | 2
  Treatment-related TEAE | 2 | 1
  All-causality SAE | 0 | 0

28. Secondary Outcome: Number of Participants With Laboratory Test Abnormality (Without Regard to Baseline Abnormality)
Description: Laboratory tests included hematology, clinical chemistry and urinalysis. Laboratory abnormalities reported in at least 1 participant are reported in this OM.
Time Frame: Maximum of 11 weeks
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6 | 6
Participants | 1 | 0

29. Secondary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Pre-Defined Criteria
Description: Vital signs data included supine systolic and diastolic blood pressure (BP) and pulse rate. Potentially clinically significant vital signs abnormalities are defined as: systolic BP - minimum (min) absolute result <90 mmHg, maximum (max) increase or decrease from baseline ≥30 mmHg; diastolic BP - min absolute result <50 mmHg, max increase or decrease from baseline ≥20 mmHg; supine pulse rate - min absolute result <40 beat per minute (bpm), max absolute result >120 bpm. Participants with vital signs data meeting any criteria above are reported in this OM.
Time Frame: Maximum of 11 weeks
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6 | 6
Participants | 0 | 1

30. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-Defined Criteria
Description: ECG data included heart rate, PR interval, QT interval, QT Interval (Fridericia's Correction) (QTcF) and QRS complex.
  Potentially clinically significant ECG abnormalities are categorized as follows: Uncorrected QT value >500 millisecond (msec). QTcF - absolute value >450 and ≤480 msec; absolute value >480 and ≤500 msec; absolute value >500 msec; increase from baseline >30 and ≤60 msec; increase from baseline >60 msec. PR interval - max absolute value ≥300 msec; baseline value >200 msec and ≥25% increase from baseline; baseline value ≤200 msec and ≥50% increase from baseline. QRS complex - max absolute value ≥140 msec; ≥50% increase from baseline. Participants with ECG data meeting any criteria above are reported in this OM, if any.
Time Frame: Maximum of 11 weeks
Population: The safety analysis population included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Maximum of 11 weeks
Description: All TEAEs, without regard to possibility of causal relationship with the study treatment, are summarized.
Arm/Group | Period 1: [14C]PF-07081532 30 mg Oral | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: [14C]PF-07081532 30 mg Oral (N=6) | Period 2: PF-07081532 30 mg Oral + [14C]PF-07081532 100 µg IV (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hunger (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT05652647/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05652647/SAP_001.pdf